CLINICAL TRIAL: NCT01338584
Title: A Randomized Controlled Trial Study of the Efficacy of Intensive Preoperative Pelvic Floor Muscle Training to Decrease Post-prostatectomy Urinary Incontinence
Brief Title: Trial Study of the Efficacy of Intensive Preoperative Pelvic Floor Muscle Training to Decrease Post-prostatectomy Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Sau-loi NG, Advanced Practice Nurse, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW 11-046
Record Dates: First submitted 2011-04-04; First posted 2011-04-19 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Urinary Incontinence
Keywords: Pelvic floor muscle training; Post prostatectomy; Early regaining of urinary continence; Positive improvement in quality of life
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pelvic floor muscle training, post prostatectomy (Experimental): Pelvic floor muscle training will be taught on the day of admission
  Interventions: Behavioral: Pelvic floor muscle training 3 weeks before radical prostatectomy; Behavioral: Intensive preoperative pelvic floor muscle training

INTERVENTIONS:
Behavioral: Pelvic floor muscle training 3 weeks before radical prostatectomy — Participants in the intervention group need to attend the nurse-led clinic 6 times for practising pelvic floor muscle preoperatively instead of starting the exercise one day before surgery (usual management).
  Other Names: Pelvic floor muscle training
Behavioral: Intensive preoperative pelvic floor muscle training — Patient started to learn pelvic floor muscle 3 weeks before surgery
  Other Names: post prostatectomy; promote urinary continence

SUMMARY:
Urinary incontinence after radical prostatectomy is a significant clinical problem despite advances in surgical techniques. In the literature, the incidence of post prostatectomy urinary incontinence varies widely from 0.5 to 87% (Parekh et al, 2003). Various reasons are held responsible for this wide discrepancy, including surgical technique, definition of incontinence, time of evaluation, pathological stage, and patient age. The etiology of post prostatectomy urinary incontinence has been attributed to sphincteric deficiency, either from injury of striated muscle fibres or the innervating nerve fibres (Koelbl et al 2002). The effect of urinary incontinence on the quality of life in these patients has been subject to debate (Litwin et al, 1995; Braslis et al, 1995). For many patients, however, early recovery from urinary incontinence has been a major concern (Moore et al, 1999), especially in younger patients.

Various treatment modalities for post prostatectomy urinary incontinence have been introduced, including conservative managemnt such as pelvic floor muscle training, pharmacological treatment and surgical treatment. However, surgery is an invasive procedure and it's usually be the last resort. Although the Cochrane Incontinence Group (2007) commented on the need for ongoing research to clarify the role of pelvic floor muscle training, it is still the first-line treatment used to restore pelvic floor or bladder function after radical prostatectomy (MacDonald et. al., 2007). Currently, patients learned pelvic floor muscle training on the day of admission for surgery by ward staff in HA hospitals of Hong Kong. Subsequently, after removal of urethral catheter, patients will attend the nurse-led clinic for reassessment and reinforcement of pelvic floor muscle training. The continence rates which defined as zero pad were 69%, 78.7% and 88.9% at 3 months, 6 months and 12 months respectively (Tam and Ho et al., 2010). In order to determine the efficacy of intensive preoperative pelvic floor muscle training to decrease post-prostatectomy urinary incontinence, a randomized controlled trial will be conducted. Participants in the intervention group would start the pelvic floor muscle training 3 weeks before surgery provided by an urology nurse specialist whereas the control group would start the pelvic floor muscle training on the day of admission for surgery provided by ward staff. Measurement on the grams of urine loss, sense of self control in urination and quality of life are collected on 4, 8, 12 and 24 weeks after surgery for comparison between the two groups.

DETAILED DESCRIPTION:
Prostate cancer is one of the most important health problems in men. According to the information from Centre of Health Promotion (CHP) in January 2010, prostate cancer recorded the largest increase in incidence rate among the common male cancers in Hong Kong during the past two decades. In 2007, prostate cancer was the fourth most common cancer in men and there were 1 205 newly diagnosed cases of prostate cancer. It accounted for 9.2% of all new cancer cases in males. It is the fifth leading cause of male cancer deaths in Hong Kong. In 2008, a total of 282 men died from this cancer, accounting for 3.8% of male cancer deaths.

For patients with disease confined to the prostate, several treatment alternatives are now available. However, radical prostatectomy remains the standard for long-term cure (Guidelines of American Urological Association, 2010). The incidence of incontinence and erectile dysfunction is higher after operation than other therapies for localized prostate cancer (Alivizatos, et al, 2005). Based on the literature review, the post prostatectomy urinary incontinence (PPUI) rates were ranging from 0.5-87% (Parekh, et al, 2003) and potency rates ranging from 11-87% (Alivizatos, et al, 2005). Various reasons are held responsible for this wide discrepancy, including surgical technique, definition of incontinence, time of evaluation, pathological stage, and patient age (Pannek & Konig, 2005). However, the majority of the patients undergoing radical prostatectomy would vote for the operation again as they put tumour free on their first priority (Alivizatos, et al., 2005). The cause of urinary incontinence after radical prostatectomy is not completely understood, but leakage is thought to result primarily from sphincteric insufficiency, resulting from sphincteric injury or detrusor overactivity and effects on the bladder detrusor muscle (Leach, 1995). Men afflicted with urinary incontinence must contend with shame, embarrassment, depression, avoidance of social activities and altered life style (Braslis et al., 1995; Herr, 1994). So, early and appropriate management of urinary incontinence can improve one's quality of life and reduce the adverse consequences of urinary incontinence such as lowering of the physical health causing disability and dependence, affecting the psychological well-being and social functioning; as well as escalating health care costs (White & Getliffe, 2003; Wyman, 2003).

Sueppel et al. (2001) found that pelvic floor muscle training (PFMT) taught pre operatively helped patients achieve continence quicker than if only taught post operatively. There was significant improvement in the intervention group objectively by weighting the pad in every visit (pad weight: 2.8 g in intervention group whereas 33.3 g in control group). Previously, Bales et al. (2000) recruited 100 men scheduled to undergo radical prostatectomy were randomized to receive PFMT with biofeedback 2-4 weeks before surgery by a nurse pre and post operatively or to a group only receive briefly verbal instruction on PFMT without biofeedback. Six months following surgery, the continence rates, as defined by the use of one pad or less per day were 96% (44 of 47) and 96% (48 of 50) in the biofeedback and control groups respectively. The authors concluded that pre operative formal PFMT and biofeedback training did not improve the outcome of PFMT on overall continence as measured by number of pads used or the rate of return of urinary control in men undergoing radical prostatectomy at 6 months (p=0.596).

Among all studies reviewed, the efficacy of pre operative PFMT in early regaining of urinary control after radical prostatectomy is still inconclusive. Thus, further studies on PFMT for PPUI are needed (Centemero & Rigatti, et al., 2010).

ELIGIBILITY:
Inclusion Criteria:

* Chinese;
* Physically able to complete the pad test

Exclusion Criteria:

* Prior bladder surgery;
* Prior urinary incontinence;
* Neurogenic dysfunction of the lower urinary tract;
* Pre-operative history of overactive bladder;
* Impaired mental status;
* Allergic to latex.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change in grams of urine loss at different intervals post surgery | 4, 8, 12, and 24 weeks post surgery
  To determine the benefit of starting intensive PFMT before radical prostatectomy and continuing PFMT postoperatively in order to promote (1) early regaining of urinary continence in the intervention group by weighted pad after pad test and (2) any positive improvement in quality of life in the intervention group.

SECONDARY OUTCOMES:
Change in patients' sense of self control in urination and quality of life at different intervals post surgery | 4, 8, 12, and 24 weeks post surgery
  1. The intervention group will significantly regain bladder control by decreasing urine leakage as measured by pad test than the control group by the end of three months post surgery.
  2. The intervention group will report better quality of life as measured by the Functional Assessment of Cancer Therapy-Prostate (FACT-P), Incontinence Impact on Quality (IIQ-7) and Health-related Quality of Life (SF 12)

CONTACTS AND LOCATIONS:
Overall Officials: Sau-loi NG, Principal Investigator — The University of Hong Kong & Queen Mary Hospital
Locations (1):
- NG Sau-loi, Hong Kong, Heng Fa Chuen, Hong Kong

REFERENCES:
- [Background] Hunter KF, Moore KN, Glazener CM. Pelvic floor muscle training to improve urinary incontinence after radical prostatectomy: a systematic review of effectiveness. BJU Int. 2007 Nov;100(5):1191; author reply 1191-2. doi: 10.1111/j.1464-410X.2007.07248_1.x. No abstract available. PMID 17922792
- [Background] Novara G. Editorial comment on: does physiotherapist-guided pelvic floor muscle training reduce urinary incontinence after radical prostatectomy? A randomised clinical trial. Eur Urol. 2008 Aug;54(2):447. doi: 10.1016/j.eururo.2008.04.023. Epub 2008 Apr 18. No abstract available. PMID 18448232
- See also: The University of Hong Kong — http://hku.hk